CLINICAL TRIAL: NCT00550121
Title: Does Ascorbic Acid Reduce Sympathoexcitation in CHF?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CHFVIT
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: vitamin C
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin C
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
In CHF central sympathetic activity is increased. ROS formation seems to play a role in this process. This study analyzes the effect of vitamin C as an antioxidant on central sympathetic activity in CHF

ELIGIBILITY:
Inclusion Criteria:

* Heart failure of at least New York Heart Association (NYHA) class II
* Left ventricular ejection fraction (LVEF) <= 40%
* Age 20-80 years

Exclusion Criteria:

* Necessity of short-term PCI, CABG or heart transplantation,
* Chronic disease of the autonomic nervous system,
* diabetes mellitus,
* use of tricyclic antidepressant drugs and/or a-adrenergic receptor antagonists.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-08; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
change in central sympathetic output after vitamin C vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Cees J Tack, MD, PhD, Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands